CLINICAL TRIAL: NCT03860207
Title: Phase I/II Study of Humanized 3F8 Bispecific Antibody (Hu3F8-BsAb) in Patients With Relapsed/Refractory Neuroblastoma, Osteosarcoma, and Other GD2(+) Solid Tumors
Brief Title: Study of the Safety and Efficacy of Humanized 3F8 Bispecific Antibody (Hu3F8-BsAb) in Patients With Relapsed/Refractory Neuroblastoma, Osteosarcoma and Other Solid Tumor Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: study terminated due to business priorities
Sponsor: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-034
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Neuroblastoma; Osteosarcoma; Other Solid Tumor Cancers
Keywords: Humanized 3F8 Bispecific Antibody (Hu3F8-BsAb); 18-034
MeSH Terms: conditions — Neuroblastoma; Osteosarcoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This phase I/II trial will assess the toxicity and pharmacokinetics (PK) of the humanized anti-GD2 x anti-CD3 bispecific antibody (hu3F8-BsAb) in phase I and the anti-tumor activity of hu3F8-BsAb in phase II.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hu3F8-BsAb (Experimental): Phase I Hu3F8-BsAb is given IV over ~1-3 hours on Days 1 and 8 for each cycle. In cycle 1, blood is drawn for PK studies.Phase II Hu3F8-BsAb is given IV over ~1-3 hours on Days 1 and 8 for each cycle.
  Interventions: Biological: Humanized 3F8 Bispecific Antibody; Other: Blood draw

INTERVENTIONS:
Biological: Humanized 3F8 Bispecific Antibody — Phase I Hu3F8-BsAb is given IV over ~1-3 hours on Days 1 and 8 for each cycle.Phase II Hu3F8-BsAb is given IV over ~1-3 hours on Days 1 and 8 for each cycle.
  Other Names: Humanized 3F8 Bispecific Antibody (Hu3F8-BsAb)
Other: Blood draw — In cycle 1, blood is drawn for PK studies.

SUMMARY:
The purpose of this study is to test the safety of a study drug called humanized 3F8 bispecific antibody (Hu3F8-BsAb).

ELIGIBILITY:
Inclusion Criteria:

Phase I

* Patients must have either (1) a diagnosis of NB as defined by international criteria,i.e.,histopathology (confirmed by the MSKCC Department of Pathology) or BM metastases plus high urine catecholamine levels, or (2) high grade osteosarcoma verified by histopathology (confirmed by the MSKCC Department of Pathology), or (3) other GD2-expressing solid tumor.
* For tumors other than NB and osteosarcoma, only tumors known to be GD2 positive are eligible: melanoma, desmoplastic small round cell tumors, retinoblastoma, medulloblastoma, and soft tissue sarcomas including liposarcoma, fibrosarcoma, malignant fibrous histiocytoma, leiomyosarcoma, and spindle cell sarcoma. Patients with medulloblastoma are eligible only if they have metastatic disease outside the CNS (e.g. in the bone marrow)
* NB patients must have chemorefractory (e.g. refractory to standard induction chemotherapy including cyclophosphamide, vincristine, cisplatin, etoposide) or relapsed high-risk (HR) neuroblastoma. HR NB is defined as MYCN-amplified stage 3/4/4S of any age, or MYCNnonamplified stage 4 in patients > 18 months of age at diagnosis.
* Osteosarcoma patients must have relapsed or refractory osteosarcoma after receiving standard systemic chemotherapy (e.g. combination methotrexate, doxorubicin, and cisplatin [MAP]).
* For non-NB and non-osteosarcoma tumors known to be GD2(+), patients must have relapsed or refractory disease that is resistant to standard therapy.

Phase II

Group 1:

* NB patients must have chemo refractory or relapsed HR NB. HR NB is defined as MYCNamplified stage 3/4/4S of any age, or MYCN-nonamplified stage 4 in patients > 18 months of age at diagnosis.
* The diagnosis of NB must be defined by international criteria i.e., histopathology (confirmed by the MSKCC Department of Pathology) or BM metastases plus high urine catecholamine levels.

Group 2:

* Patients must have a diagnosis of high grade osteosarcoma defined by histopathology (confirmed by the MSKCC Department of Pathology).
* Patients must have relapsed or refractory osteosarcoma after receiving standard systemic chemotherapy (e.g. combination methotrexate, doxorubicin, and cisplatin [MAP]).

All criteria below are common to both phase I and phase II:

Disease status

* For NB patients, patients must have measurable or evaluable disease (e.g. abnormal findings in computed tomography (CT), magnetic resonance imaging (MRI), metaiodobenzylguanidine (MIBG) scan, or positron emission tomography (PET)) OR morphologic evidence of disease in bone marrow.
* For osteosarcoma or other GD2(+) solid tumor patients, patients must have measurable disease.

Other criteria:

* Patients must be ≥ 1 year of age ( protocol amendment 1.0-5.0)
* Patients must be ≥ 1 year of age and < 18 years of age (protocol amendment 6.0-10.0)
* Patients with prior exposure to anti-GD2 antibodies must have a negative HAHA antibody titer
* Adequate hematopoietic function defined as:

  * Absolute neutrophil count ≥500/ul
  * Absolute lymphocyte count ≥500/ul
  * Platelet count ≥25,000/ul
* Negative serum pregnancy test in women of child-bearing potential.
* Women of child-bearing potential must be willing to practice an effective method of birth control while on treatment.
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Patients who are in complete remission.
* Existing severe major organ dysfunction. i.e. renal, cardiac, hepatic, neurologic, pulmonary, or gastrointestinal toxicity ≥ Grade 3 except for hearing loss, alopecia, anorexia, nausea, hyperbilirubinemia or hypomagnesemia from TPN, which may be Grade 3.
* Hematologic and active CNS malignancies including CNS metastasis.
* Active life-threatening infection.
* Pregnant women or women who are breast-feeding.
* Inability to comply with protocol requirements.
* History of autoimmune disease with potential CNS involvement or a current autoimmune disease.
* Chemotherapy or immunotherapy within three weeks prior to study enrollment. T-cell based immunotherapies (e.g. CAR-modified T cells, checkpoint inhibitors) should have been completed >6 weeks prior to treatment with hu3F8-BsAb.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.009 mcg/kg/Cycle: Dose Level 1 (0.009 mcg/kg/cycle) is the starting dose Phase I Hu3F8-BsAb Dose level 1 (0.009 mcg/kg/cycle) is given IV over ~1-3 hours on Days 1 (0.0045 mcg/kg) and 8 (0.0045 mcg/kg) for each cycle.
- 0.09 mcg/kg/Cycle: Phase I Hu3F8-BsAb Dose level 2 (0.09 mcg/kg/cycle) is given IV over ~1-3 hours on Days 1 (0.045 mcg/kg) and 8 (0.045 mcg/kg) for each cycle.
- 0.9 mcg/kg/Cycle: Phase I Hu3F8-BsAb Dose level 3 (0.9 mcg/kg/cycle) is given IV over ~1-3 hours on Days 1 (0.45 mcg/kg) and 8 (0.45 mcg/kg) for each cycle.
- 2.6 mcg/kg/Cycle: Phase I Hu3F8-BsAb Dose level 4 (2.6 mcg/kg/cycle) is given IV over ~1-3 hours on Days 1 (1.3 mcg/kg) and 8 (1.3 mcg/kg) for each cycle.
- 4.8 mcg/kg/Cycle: Phase I Hu3F8-BsAb Dose level 5 (4.8 mcg/kg/cycle) is given IV over ~1-3 hours on Days 1 (1.3 mcg/kg) and 8 (3.5 mcg/kg) for each cycle.
- 9.3 mcg/kg/Cycle: Phase I Hu3F8-BsAb Dose level 6 (9.3 mcg/kg/cycle) is given IV over ~1-3 hours on Days 1 (1.3 mcg/kg) and 8 (8 mcg/kg) for each cycle.
Period: Overall Study
Arm/Group | 0.009 mcg/kg/Cycle | 0.09 mcg/kg/Cycle | 0.9 mcg/kg/Cycle | 2.6 mcg/kg/Cycle | 4.8 mcg/kg/Cycle | 9.3 mcg/kg/Cycle
Started | 1 | 1 | 1 | 3 | 2 | 3
Safety Analysis Set | 1 | 1 | 1 | 3 | 2 | 3
Discontinued the Treatment | 1 | 1 | 1 | 3 | 2 | 3
Discontinued Treatment - Adverse Events | 0 | 0 | 0 | 0 | 0 | 2
Discontinued Treatment - Progressive Disease | 1 | 1 | 1 | 3 | 2 | 1
Completed (Completed minimum 30 days of follow-up from end of treatment.) | 1 | 1 | 1 | 2 | 2 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set.
  In Protocol version 1.0 to 5.0 patients ≥ 1 year were eligible. In Protocol version 6.0 to 10.0 patients between ≥ 1 year and < 18 years were eligible.
Groups:
- 0.009 mcg/kg/Cycle: Phase I Hu3F8-BsAb Dose level 1 (0.009 mcg/kg/cycle) is given IV over ~1-3 hours on Days 1 (0.0045 mcg/kg) and 8 (0.0045 mcg/kg) for each cycle.
- 0.09 mcg/kg/Cycle: Phase I Hu3F8-BsAb Dose level 2 (0.09 mcg/kg/cycle) is given IV over ~1-3 hours on Days 1 (0.045 mcg/kg) and 8 (0.45 mcg/kg) for each cycle.
- Total: Total of all reporting groups
Arm/Group | 0.009 mcg/kg/Cycle | 0.09 mcg/kg/Cycle | 0.9 mcg/kg/Cycle | 2.6 mcg/kg/Cycle | 4.8 mcg/kg/Cycle | 9.3 mcg/kg/Cycle | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 2 | 3 | 11
Age, Customized [Count of Participants; unit: Participants]
  0- 6 years | 1 | 0 | 0 | 1 | 0 | 0 | 2
  7-11 years | 0 | 1 | 1 | 1 | 1 | 0 | 4
  12-17 years | 0 | 0 | 0 | 0 | 0 | 1 | 1
  18 years and above | 0 | 0 | 0 | 1 | 1 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 3 | 0 | 0 | 4
  Male | 1 | 1 | 0 | 0 | 2 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 1 | 3 | 2 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 1 | 1 | 1 | 2 | 1 | 3 | 9
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 3 | 2 | 3 | 11
Disease Type [Count of Participants; unit: Participants]
  High Grade Ostersarcoma | 0 | 0 | 0 | 1 | 1 | 2 | 4
  Neuroblastoma | 1 | 1 | 1 | 2 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLTs) Phase I
Description: Summary of DLTs in DLT evaluable subjects.
Time Frame: Days 1 through 28 in cycle 1
Population: DLT Evaluable Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | 0.009 mcg/kg/Cycle | 0.09 mcg/kg/Cycle | 0.9 mcg/kg/Cycle | 2.6 mcg/kg/Cycle | 4.8 mcg/kg/Cycle | 9.3 mcg/kg/Cycle
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 2 | 3
Participants
  Any DLT | 0 | 0 | 0 | 0 | 0 | 2
  DLT Type - Nervous system disorder: number analyzed (Participants) | 0 | 1 | 1 | 3 | 2 | 3
  DLT Type - Nervous system disorder | 0 | 0 | 0 | 0 | 0 | 1
  DLT Type - Syncope | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From 1st dose to 30 days after last dose
Description: The table shows TEAEs with onset prior to 31 days after last dose of Hu3F8-BsAb.
  Treatment Emergent Adverse Event are either events with start date and time after initiation of treatment, or event that may have worsened on or after initiation of treatment. No patients experienced fatal AEs
Arm/Group | 0.009 mcg/kg/Cycle | 0.09 mcg/kg/Cycle | 0.9 mcg/kg/Cycle | 2.6 mcg/kg/Cycle | 4.8 mcg/kg/Cycle | 9.3 mcg/kg/Cycle
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 1/1 | 2/3 | 2/2 | 3/3
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 0/1 | 1/3 | 1/2 | 3/3
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 3/3 | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.009 mcg/kg/Cycle (N=1) | 0.09 mcg/kg/Cycle (N=1) | 0.9 mcg/kg/Cycle (N=1) | 2.6 mcg/kg/Cycle (N=3) | 4.8 mcg/kg/Cycle (N=2) | 9.3 mcg/kg/Cycle (N=3)
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.009 mcg/kg/Cycle (N=1) | 0.09 mcg/kg/Cycle (N=1) | 0.9 mcg/kg/Cycle (N=1) | 2.6 mcg/kg/Cycle (N=3) | 4.8 mcg/kg/Cycle (N=2) | 9.3 mcg/kg/Cycle (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 2 | 3
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 1 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pupils unequal (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 2
Chills (General disorders) | 0 | 0 | 0 | 1 | 1 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 2 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 2 | 1 | 2
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 2 | 2 | 3
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 1 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 1 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 3 | 2 | 1
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Haemoglobin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2
Lymphocyte count decreased (Investigations) | 1 | 1 | 1 | 3 | 2 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 3 | 2 | 2
Platelet count decreased (Investigations) | 0 | 1 | 1 | 2 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 1 | 1 | 2 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 1 | 0 | 2 | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 2 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 2 | 3

LIMITATIONS AND CAVEATS:
The study was terminated after 11 subjects due to a business strategy decision. At this point the maximum tolerated dose was not established.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT03860207/Prot_002.pdf
  • Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT03860207/SAP_003.pdf